CLINICAL TRIAL: NCT00780858
Title: GnRH Antagonist Prevention of Premature Luteinization in Patients Undergoing IUI
Brief Title: Premature Luteinization Prevention by GnRH Antagonist in Patients Undergoing IUI
Acronym: LP
Status: Completed | Type: Observational
Sponsor: IVI Madrid (Other)
Responsible Party: Principal Investigator, Juan A Garcia-Velasco, MD, IVI Madrid
Other Study IDs: IVIMAD-JMS-09-2008-02
Record Dates: First submitted 2008-10-25; First posted 2008-10-28 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Infertility
Keywords: GnRH antagonist; IUI
MeSH Terms: conditions — Infertility | interventions — ganirelix

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Ganirelix: Patients with premature lutenization (progesterone >1,2 ng/ml) who did not get pregnant during the first IUI underwent a second IUI.
  Interventions: Drug: Ganirelix
- Control: Patients without premature lutenization (progesterone >1,2 ng/ml) underwent a only one IUI.

INTERVENTIONS:
Drug: Ganirelix — Ganirelix 0.25mg s.c every 24 h starting stimulation day 6
  Other Names: Orgalutran
  Groups: Ganirelix

SUMMARY:
Premature luteinization in patients undergoing IUI can occur in up to 24% of cycles. These patients, according to recent data, have a lower pregnancy rate than controls. The possibility to avoid premature luteinization with GnRH antagonist may restore the chances of achieving a pregnancy in these women.

DETAILED DESCRIPTION:
The purpose of this study was to investigate whether a subset of patients benefits from GnRHa administration during IUI. PL was tested for in patients who were undergoing artificial insemination procedures, and the effect of GnRHa on PR in patients who

ELIGIBILITY:
Inclusion Criteria:

* previous failed IUI cycle with premature luteinization

Exclusion Criteria:

* 39 years or older
* not eligible for IUI (patent tubes, > 3 million capacitated spermatozoa)
* 4 previous IUI cycles

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Healthy women with patent tubes who were undergoing IUI due to infertily of unknown origin.
Sampling Method: Non-Probability Sample
Enrollment: 662 (Actual)
Dates: Start 2008-10; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate | 2 weeks after intervention

SECONDARY OUTCOMES:
premature luteinization | at the time of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Juan antonio García-Velasco, MD, Principal Investigator — IVI Madrid
Locations (1):
- IVI-Madrid, Madrid, Spain

REFERENCES:
- [Background] Kosmas IP, Tatsioni A, Kolibianakis EM, Verpoest W, Tournaye H, Van der Elst J, Devroey P. Effects and clinical significance of GnRH antagonist administration for IUI timing in FSH superovulated cycles: a meta-analysis. Fertil Steril. 2008 Aug;90(2):367-72. doi: 10.1016/j.fertnstert.2007.06.064. Epub 2007 Oct 23. PMID 17936285